CLINICAL TRIAL: NCT03219476
Title: Neoadjuvant Endocrine Therapy in Hormone Receptor-Positive HER2-Negative Node-Negative Breast Cancer Patients to Assess Responses and Mechanisms of Endocrine Resistance
Brief Title: Neoadjuvant Endocrine Therapy in Hormone Receptor-Positive, Human Epidermal Growth Factor Receptor 2 (HER2)-Negative Node-Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Lubna Chaudhary, Associate Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO30178
Record Dates: First submitted 2017-07-12; First posted 2017-07-17 (Actual); Results first posted 2022-10-18 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer; Invasive Breast Cancer
Keywords: aromatase inhibitor; breast cancer; estrogen receptor; progesterone receptor; endocrine-targeted therapy; Anti-estrogen therapy; HR+; HER2-negative; Neoadjuvant Treatment
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole; Letrozole; exemestane; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neoadjuvant endocrine therapy treatment (physician's choice) (Experimental): Once enrolled, patients would be treated with the current standard-of-care endocrine therapy. Choice of endocrine therapy (aromatase inhibitors or tamoxifen) would be decided by medical oncologist, following a review of the patient's medical history and menstrual status. The patient would be treated with endocrine therapy in a neoadjuvant setting for four weeks, with dosing continuing until surgery.
  Interventions: Drug: Anastrozole; Drug: Letrozole; Drug: Exemestane; Drug: Tamoxifen

INTERVENTIONS:
Drug: Anastrozole — 1 mg once daily.
  Other Names: Arimidex
Drug: Letrozole — 2.5mg once daily.
  Other Names: Femara
Drug: Exemestane — 25 mg once daily.
  Other Names: Aromasin
Drug: Tamoxifen — 20 mg once daily.
  Other Names: Soltamox

SUMMARY:
This is an exploratory interventional study that initiates standard-of-care anti-estrogen treatment preoperatively for four weeks.

DETAILED DESCRIPTION:
STUDY RATIONALE: Patients with hormone receptor (HR)+, HER2- node-negative breast cancers generally undergo surgical resection upfront, followed by adjuvant chemotherapy, if needed, in addition to adjuvant endocrine therapy. Because endocrine therapy is primarily delivered in the postoperative setting, the ability to assess the tumor response to this treatment modality is lost and very difficult to assess. This study offers the unique opportunity to assess the responsiveness of breast tumors to endocrine therapy while the tumors are still in vivo by treating patients with endocrine therapy before surgery and assessing molecular changes with treatment. By comparing pre- and post-treatment levels of molecular markers in individual tumors, the team expects to identify predictors of responsiveness to existing agents and identify new candidate therapeutic targets.

PRIMARY OBJECTIVE: The primary objective is to determine the frequency of increased HER family of receptor tyrosine kinases protein expression in tumors, following treatment with neoadjuvant endocrine therapy and their correlation with Ki-67 tumor responses. The team will measure cancer cell protein levels of growth factor receptors of the human epidermal growth factor receptor (HER) family before and after neoadjuvant endocrine therapy. The data will be used to inform a future randomized trial of combined endocrine and the most promising anti-HER targeted therapy.

ELIGIBILITY:
Inclusion Criteria:

* Female; age ≥18 years.
* Pathologically proven diagnosis of invasive breast cancer, clinically stage I-II.
* Clinically lymph node negative, confirmed by clinical exam and/or ultrasound imaging.
* Estrogen- and/or progesterone-receptor-positive tumor, defined ≥1% positively staining cells by immunohistochemistry, according to the current American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines.
* HER2/neu must be negative by immunohistochemistry (IHC) or fluorescence in situ hybridization (FISH).
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Pretreatment evaluations (minimum diagnostic workup) within 28 days prior to study
* Qualify for anti-endocrine treatment (per medical oncologist).
* Informed consent provided.
* If history of contralateral breast cancer, patient completed all treatment two years prior
* No treatment for this breast cancer or any malignancy within two years (except non-melanomatous skin cancer, carcinoma in situ of the cervix and contralateral breast cancer)
* Using adequate methods of contraception; negative pregnancy test.
* No strong CYP2D6 inhibitors.
* Adequate organ function with baseline lab values.

  * Absolute neutrophil count (ANC) ≥ 1500/µL.
  * Hemoglobin (Hb) ≥ 9g/dL.
  * Platelet count ≥ 100,000/µL.
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3x upper limit of normal (ULN).
  * Serum bilirubin within ≤ 1.5 x ULN.

Exclusion Criteria:

* American Joint Committee on Cancer (AJCC) clinical T4, N1-3 or M1, breast cancer.
* Synchronous non-breast malignancy (exceptions include non-melanomatous skin cancer, carcinoma in situ of the cervix).
* Purely noninvasive breast cancer (i.e., ductal carcinoma in situ, lobular carcinoma in situ).
* Men with breast cancer.
* Medical, psychiatric or other condition that would prevent the patient from receiving the protocol therapy or providing informed consent.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Cis females.
Enrollment: 37 (Actual)
Dates: Start 2017-02-05 (Actual); Primary Completion 2020-02-04 (Actual); Study Completion 2025-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lubna Chaudhary, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chaudhary LN, Jorns JM, Sun Y, Cheng YC, Kamaraju S, Burfeind J, Gonyo MB, Kong AL, Patten C, Yen T, Cortina CS, Carson E, Johnson N, Bergom C, Tsaih SW, Banerjee A, Wang Y, Chervoneva I, Weil E, Chitambar CR, Rui H. Frequent upregulation of HER2 protein in hormone-receptor-positive HER2-negative breast cancer after short-term neoadjuvant endocrine therapy. Breast Cancer Res Treat. 2023 Oct;201(3):387-396. doi: 10.1007/s10549-023-07038-3. Epub 2023 Jul 17. PMID 37460683

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Neoadjuvant Endocrine Therapy Treatment (Physician's Choice)
Started | 37
Completed | 37
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Neoadjuvant Endocrine Therapy Treatment (Physician's Choice)
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 36
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Change in Baseline of Cancer Cell Protein Levels of Human Epidermal Growth Factor Receptor (HER) Family Members (HER1-4) Following Neoadjuvant Endocrine Therapy.
Description: ImmunoHistoChemistry (IHC) will be used. The IHC test gives a score of 0 to 3+ that measures the amount of HER2 receptor protein on the surface of cells in a breast cancer tissue sample. If the score is 0 to 1+ (up to 25% of cells stained), it's called "HER2 negative." If the score is 2+ (approximately 50% of cells stained), it's called "borderline." A score of 3+ (approximately 75% or more of cells stained) is called "HER2 positive." Upregulation means increased staining from a prior observation; Downregulation means decreased staining from a prior observation; and No Change means similar staining from a prior observation.
Time Frame: At four weeks.
Population: All 37 subjects were analyzed for each of the protein markers.
Measure: Count of Participants; unit: Participants
Groups:
- Change From Baseline in Human Epidermal Growth Factor Receptor 1 (HER1) Cell Protein Levels.: ImmunoHistoChemistry (IHC) will be used. The IHC test gives a score of 0 to 3+ that measures the amount of Human Epidermal Growth Factor Receptor 1 (HER1) receptor protein on the surface of cells in a breast cancer tissue sample. If the score is 0 to 1+, it's called "HER1 negative." If the score is 2+, it's called "borderline." A score of 3+ is called "HER1 positive."
- Change From Baseline in Human Epidermal Growth Factor Receptor 2 (HER2) Cell Protein Levels.: ImmunoHistoChemistry (IHC) will be used. The IHC test gives a score of 0 to 3+ that measures the amount of Human Epidermal Growth Factor Receptor 2 (HER2) receptor protein on the surface of cells in a breast cancer tissue sample. If the score is 0 to 1+, it's called "HER2 negative." If the score is 2+, it's called "borderline." A score of 3+ is called "HER2 positive."
- Change From Baseline in Human Epidermal Growth Factor Receptor 3 (HER3) Cell Protein Levels.: ImmunoHistoChemistry (IHC) will be used. The IHC test gives a score of 0 to 3+ that measures the amount of Human Epidermal Growth Factor Receptor 3 (HER3) receptor protein on the surface of cells in a breast cancer tissue sample. If the score is 0 to 1+, it's called "HER3 negative." If the score is 2+, it's called "borderline." A score of 3+ is called "HER3 positive."
- Change From Baseline in Human Epidermal Growth Factor Receptor 4 (HER4) Cell Protein Levels.: ImmunoHistoChemistry (IHC) will be used. The IHC test gives a score of 0 to 3+ that measures the amount of Human Epidermal Growth Factor Receptor 4 (HER4) receptor protein on the surface of cells in a breast cancer tissue sample. If the score is 0 to 1+, it's called "HER4 negative." If the score is 2+, it's called "borderline." A score of 3+ is called "HER4 positive."
Arm/Group | Change From Baseline in Human Epidermal Growth Factor Receptor 1 (HER1) Cell Protein Levels. | Change From Baseline in Human Epidermal Growth Factor Receptor 2 (HER2) Cell Protein Levels. | Change From Baseline in Human Epidermal Growth Factor Receptor 3 (HER3) Cell Protein Levels. | Change From Baseline in Human Epidermal Growth Factor Receptor 4 (HER4) Cell Protein Levels.
Number analyzed (Participants) | 37 | 37 | 37 | 37
Participants
  Upregulation | 1 | 17 | 1 | 1
  Downregulation | 0 | 2 | 18 | 18
  No Change | 36 | 18 | 18 | 18

2. Secondary Outcome: Number of Subjects Who Achieve Complete Radiographic Response.
Description: This will be assessed by World Health Organization (WHO) criteria:
  * Complete Response (CR): The disappearance of all known disease, based on a comparison between the measurements at baseline and after four weeks of treatment with neoadjuvant therapy.
  * Partial Response (PR): A 50% or greater decrease in the product of the bi-dimensional measurements of the lesion (total tumor size), based on a comparison between the measurements at baseline and after four weeks of treatment with neoadjuvant therapy.
  * No Change (NC): A 50% decrease in total tumor size cannot be established nor has a 25% increase in the size of the lesion been demonstrated.
  * Progressive Disease (PD): A 25% or greater increase in the total tumor size of the measurable lesions (calculated on the smallest diameter recorded over time).
Time Frame: At four weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant Endocrine Therapy Treatment (Physician's Choice)
Number analyzed (Participants) | 37
Participants | 0

3. Secondary Outcome: Number of Subjects Who Achieve a Partial Radiographic Response.
Description: as for outcome 2
Time Frame: At four weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant Endocrine Therapy Treatment (Physician's Choice)
Number analyzed (Participants) | 37
Participants | 1

ADVERSE EVENTS:
Time Frame: Four weeks.
Arm/Group | Neoadjuvant Endocrine Therapy Treatment (Physician's Choice)
All-Cause Mortality (participants affected / at risk) | 1/37
Serious Adverse Events (participants affected / at risk) | 1/37
Other Adverse Events (participants affected / at risk) | 2/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neoadjuvant Endocrine Therapy Treatment (Physician's Choice) (N=37)
Infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neoadjuvant Endocrine Therapy Treatment (Physician's Choice) (N=37)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-11-27): https://cdn.clinicaltrials.gov/large-docs/76/NCT03219476/Prot_SAP_000.pdf
  • Informed Consent Form (2019-01-09): https://cdn.clinicaltrials.gov/large-docs/76/NCT03219476/ICF_001.pdf